CLINICAL TRIAL: NCT03842462
Title: NHFOV vs NIPPV vs nCPAP in Preterm Infants With Respiratory Distress Syndrome: A Multi-center, Prospective, Randomized, Controlled Clinical Superior Trial
Brief Title: NHFOV vs NIPPV vs nCPAP in Preterm Infants With Respiratory Distress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiulongpo No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, Xingwang Zhu, Doctor, Jiulongpo No.1 People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHFOV study group
Record Dates: First submitted 2019-01-31; First posted 2019-02-15 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Preterm Infant
Keywords: Preterm Infant; Respiratory distress syndrome; nasal continuous positive airway pressure; noninvasive intermittent positive airway pressure; noninvasive high-frequency oscillatory ventilation
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nCPAP (Active Comparator): neonates assigned to the nCPAP group will be started on a pressure of 6 cmH2O( adjust range:6-8 cmH2O) by pure CPAP system , with FiO2 (0.21～0.40)adjusted to target SpO2 from 89% to 94%
  Interventions: Other: nCPAP
- NIPPV (Active Comparator): neonates assigned to the NIPPV group will be started with the following parameters: a) positive end-expiratory pressure (PEEP) of 4 cmH2O (can be raised in steps of 1 cmH2O to max 8 cmH2O, according to the oxygenation).b)Peak Inspiratory Pressure (PIP) of15 cmH2O (can be raised in steps of 1 cmH2O to max 25 cmH2O, according to oxygenation,PaCO2 levels and the chest expansion); maximal allowed FiO2 will be 0.40 and SpO2 targets will be 90-95%. c) inspiratory time (IT) will be 0.45 - 0.5 sec (according to clinicians'evaluation of leaks and the appearance of the pressure curve: a small pressure plateau is required and flow may be set accordingly) and rate will be started at30 bpm (can be raised in steps of 5 bpm to max 50 bpm, according to PaCO2 levels).
  Interventions: Other: NIPPV
- NHFOV (Experimental): - neonates assigned to NHFOV will be started with the following boundaries, according to available physiological and mechanical data, as suggested elsewhere:
  a) Paw of 10 cmH2O (can be changed in steps of 1 cmH2O within the range range 5- 16cmH2O); Paw will be titrated (within the range) according to open lung strategy, performing alveolar recruitment. Maximal allowed FiO2 will be 0.40 and SpO2 targets will be 89%-94%. b) frequency of 10Hz(can be changed in steps of 1Hz within the range 8-15Hz). c)Inspiratory time 50% (1:1).[ d)amplitude 25 cmH2O(can be changed in steps of 5 cmH2O within the range 25-50 cmH2O); amplitude will be titrated according to PaCO2.
  Interventions: Other: NHFOV

INTERVENTIONS:
Other: nCPAP — infants receive primary non-invasive respiratory support by mean of nCPAP
  Arms: nCPAP
Other: NIPPV — infants receive primary non-invasive respiratory support by mean of NIPPV
  Arms: NIPPV
Other: NHFOV — infants receive primary non-invasive respiratory support by mean of NHFOV
  Arms: NHFOV

SUMMARY:
This will be a prospective, multi-center, three-arms,parallel, randomized, controlled trial with a superiority design,conducted in China. The investigators conduct this multi-centre, randomized, controlled trial to test the hypothesis that NHFOV is more effective than nCPAP or NIPPV in the treatment of respiratory distress syndrome (RDS) in infants with a gestational age of less than 30 weeks or a birth weight of less than 1500g when used as a primary noninvasive ventilation (NIV) mode.

DETAILED DESCRIPTION:
Preterm infants are eligible to the study if they they match the following inclusion criteria: (1) Gestational age (GA) less than 30 weeks or Birth weight less than 1500g; (2) They have a diagnose of RDS, and RDS Silverman score﹥5; (3) Informed parental consent has been obtained.

Neonates will be randomized and assigned either to nCPAP, NIPPV or NHFOV arms with a 1:1:1 ratio, when patients fulfill all inclusion criteria. Randomization cannot be done earlier. Simple randomization will be done according to a computer-generated random number table and will be posted in a specific secured website 24/7 available. Twins will be allocated in the same treatment group. Infants randomized to one arm cannot crossover to the other or vice-versa during the study.

For all the groups, if the fraction of inspired oxygen (FiO2) requirement is persistently higher than 0.35-0.40 per target SpO2 89-94% and/or dyspnoea defined by Silverman score > 6 after starting the respiratory support, newborns receive Surfactant by "INSURE" technique, involving endotracheal intubation by direct laryngoscopic vision, endotracheal administration of surfactant (Curosurf, Chiesi Pharmaceutics, Parma, Italy) 200 mg/kg and finally extubation.

After the administration of surfactant, if FiO2 requirement is persistently >0.4 to keep SpO2 89-94% or severe apnea episodes are present (defined as recurrent apnea with >3 episodes/h associated with heart rate <100/min or a single episode of apnea requiring bag and mask ventilation within a 24-hour period ) or at the blood gas (arterial or free-flowing capillary blood) PaCO2>60 mmHg and potential of hydrogen (pH)<7.20 obtained at least 1 hour after commencement of the assigned treatment, newborns are intubated and mechanically ventilated. For all the newborns enrolled in the study, arterial or free-flowing capillary blood gas is checked every 6-12 hours, a cerebral and cardiac ultrasound screening is performed within 24 hrs. Further controls follow the routine of the ward.

The study intervention (nCPAP, NIPPV or NHFOV) will be stopped when the above-described minimum parameters are reached and maintained for at least 48h with the following: (1) FiO2≤0.25; (2) Silverman score <3; (3)no apneas or bradycardia without spontaneous recovery.If a baby will desaturate (SpO2<85% with FiO2>25%) or has relevant dyspnea (Silverman≧3) or more than 3 apneas/d, the intervention (CPAP, NIPPV or NHFOV) will be restarted for at least 48h and then re-evaluated

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) of less than 30 weeks or birth weight less than 1500g
* Clinical diagnose of RDS
* Parental consent

Exclusion Criteria:

* Intubated for resuscitation or for other reasons at birth
* Major congenital malformations or known complex congenital heart disease
* No parental consent

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 684 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-05-21 (Estimated); Study Completion 2022-05-21 (Estimated)

PRIMARY OUTCOMES:
treatment failure within 72 hours after randomization 72 hours after randomization | within 72 hours after randomization
  need for invasive mechanical ventilation

SECONDARY OUTCOMES:
Rate of airleaks(pneumothorax and/or pneumomediastinum) occurred during noninvasive respiratory support | during noninvasive respiratory support
  determined by the treating clinician by the treating clinician
Rate of bronchopulmonary dysplasia | 36 weeks of postmenstrual age
  defined according to the NICHD definition
Rate of retinopathy of prematurity (ROP) | Within 6 months after birth
  ≥ 2nd stage
Rate of necrotizing enterocolitis (NEC) | through study completion, an average of 1 year
  ≥ 2nd stage
Rate of intraventricular hemorrhage | through study completion, an average of 1 year
  ≥ 3nd grade

OTHER OUTCOMES:
Rate of thick secretions causing an airway obstruction. | during noninvasive respiratory support
  determined by the treating clinician by the treating clinician
days of hospitalization | through study completion, an average of 1 year
  days
duration of noninvasive respiratory support | duration of noninvasive respiratory support
  hours
days on supplemental oxygen | through study completion, an average of 1 year
  days
need for surfactant and caffeine treatment | through study completion, an average of 1 year
  determined by the treating clinician by the treating clinician
in-hospital mortality | through study completion, an average of 1 year
  Death
Rate of nasal trauma | through study completion, an average of 1 year
  determined by the treating clinician by the treating clinician

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, PhD, Study Chair — Children's Hospital of Chongqing Medical University
Locations (8):
- China (8):
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Women and Children Health Hospital, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Guiyang Maternity and Child Health Care Hospital, Guiyang, Guizhou
  - Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Hunan Children's Hospital, Changsha, Hunan
  - Chengdu Women and Children's Central Hospital, Chengdu, Sichuan
  - Kunming Children's Hospital, Kunming, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No